CLINICAL TRIAL: NCT01532765
Title: A Multicentre Randomized Clinical Trial Comparing Epiretinal Membrane Surgery With and Without Internal Limiting Membrane Peeling
Brief Title: Randomized Trial Comparing Epiretinal Membrane Surgery With and Without Internal Limiting Membrane Removal
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resident Project which was not followed through after graduation
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 422-2010
Record Dates: First submitted 2012-01-13; First posted 2012-02-14 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2015-12

CONDITIONS: Epiretinal Membrane
Keywords: Internal limiting membrane; Indocyanine green dye
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Epiretinal Membrane Surgery without ILM peel (Active Comparator)
  Interventions: Procedure: Pars plana vitrectomy and epiretinal membrane peel
- Epiretinal Membrane Surgery with ILM peel (ICG assisted) (Active Comparator)
  Interventions: Procedure: Pars plana vitrectomy and epiretinal membrane peel; Procedure: ILM peel assisted by ICG
- Combined CE & IOL and ERM surgery without ILM peel (Active Comparator)
  Interventions: Procedure: Pars plana vitrectomy and epiretinal membrane peel; Procedure: CE-IOL
- Combined CE & IOL and ERM surgery with ILM peel (ICG assisted) (Active Comparator)
  Interventions: Procedure: Pars plana vitrectomy and epiretinal membrane peel; Procedure: ILM peel assisted by ICG; Procedure: CE-IOL

INTERVENTIONS:
Procedure: Pars plana vitrectomy and epiretinal membrane peel — 23 gauge pars plana vitrectomy with diluted intravitreal triamcinolone for visualization
Procedure: ILM peel assisted by ICG — Indocyanine green dye is prepared from 25mg powder vial from AKORN INC., 10 mL diluent provided in kit. This is further diluted to final concentration of 0.5mg/mL using 50% sterile dextrose solution
  Arms: Combined CE & IOL and ERM surgery with ILM peel (ICG assisted); Epiretinal Membrane Surgery with ILM peel (ICG assisted)
Procedure: CE-IOL — Cataract extraction by phacoemulsification and insertion foldable posterior chamber intraocular lens implant
  Arms: Combined CE & IOL and ERM surgery with ILM peel (ICG assisted); Combined CE & IOL and ERM surgery without ILM peel

SUMMARY:
Macular epiretinal membrane (ERM) is a semitranslucent, avascular, fibrocellular membrane on the inner surface along the internal limiting membrane (ILM) of the retina. ERM may cause symptomatic visual disturbances and vision loss. Since the 1970s, pars plana vitrectomy has been performed to remove the membranes with few complications, and surgical results are generally good. Recurrence rates of 5-16% have been reported. Recently, ILM peeling in ERM surgery have been popularized by a number of retrospective studies and one prospective case series to minimize the rate of ERM recurrences (16% recurrence in ERM surgery with ILM peel compares to 0% recurrence in ERM surgery without ILM peel). Surgical removal of the friable and transparent ILM is difficult and increases the risk of trauma to the retina. In addition, indocyanine green (ICG), a dye commonly used intra-operatively to enhance ILM visualization, is costly and has been shown to be toxic to the retina. The investigators study will be the first randomized-controlled multi-centred clinical trial to compare the outcomes of ERM surgery with and without ILM peeling. The results will help guide and standardize the surgical treatment of macular ERM; to minimize unnecessary surgical risks, as well as to help economize healthcare cost.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* ERM on clinical exam and/or macular OCT
* Visual acuity of 20/40 or worse (attributable to ERM)

Exclusion Criteria:

* Prior surgery for ERM in the "study eye"
* Macular edema secondary to arterial/venous occlusion(s)
* Central serous retinopathy
* Age related macular degeneration
* Diabetic cystoid macular edema
* Proliferative Diabetic Retinopathy
* Uveitis

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-09; Primary Completion 2015-05 (Actual); Study Completion 2017-03-22 (Actual)

PRIMARY OUTCOMES:
Change from baseline in macular thickness on optical coherence tomography at 6 months post-surgery (intervention) | Comparing change at 6 months following surgery and baseline
Change from baseline in visual acuity at 6 months post-surgery (intervention) | Comparing change of visual acuity at 6 months following surgery and baseline

SECONDARY OUTCOMES:
Change from baseline in macular thickness on optical coherence tomography at 1 month post-surgery (intervention) | 1 month following surgery
Change from baseline in macular thickness on optical coherence tomography at 12 months post-surgery | 12 months following surgery
Change from baseline in visual acuity at 1 month post-surgery (intervention) | 1 month following surgery (intervention)
Change from baseline in visual acuity at 3 months post-surgery (intervention) | 3 months following surgery (intervention)
Change from baseline in visual acuity at 12 months post-surgery (intervention) | 12 months following surgery (intervention)
Change from baseline in visual function score based on responses to a validated visual function questionnaire (14 items) at 1 month post-surgery (intervention) | 1 month following surgery (intervention)
Change from baseline in visual function score based on responses to a validated visual function questionnaire (14 items) at 3 months post-surgery (intervention) | 3 months following surgery
Change from baseline in visual function score based on responses to a validated visual function questionnaire (14 items) at 6 months post-surgery (intervention) | 6 months following surgery
Change from baseline in visual function score based on responses to a validated visual function questionnaire (14 items) at 12 months post-surgery (intervention) | 12 months following surgery

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

REFERENCES:
- [Background] Shimada H, Nakashizuka H, Hattori T, Mori R, Mizutani Y, Yuzawa M. Double staining with brilliant blue G and double peeling for epiretinal membranes. Ophthalmology. 2009 Jul;116(7):1370-6. doi: 10.1016/j.ophtha.2009.01.024. Epub 2009 May 8. PMID 19427701
- [Background] Wise GN. Preretinal macular fibrosis. (An analysis of 90 cases). Trans Ophthalmol Soc U K (1962). 1972;92:131-40. No abstract available. PMID 4515504
- [Background] Fraser-Bell S, Ying-Lai M, Klein R, Varma R; Los Angeles Latino Eye Study. Prevalence and associations of epiretinal membranes in latinos: the Los Angeles Latino Eye Study. Invest Ophthalmol Vis Sci. 2004 Jun;45(6):1732-6. doi: 10.1167/iovs.03-1295. PMID 15161833
- [Background] Klein R, Klein BE, Wang Q, Moss SE. The epidemiology of epiretinal membranes. Trans Am Ophthalmol Soc. 1994;92:403-25; discussion 425-30. No abstract available. PMID 7886875
- [Background] Hirokawa H, Jalkh AE, Takahashi M, Takahashi M, Trempe CL, Schepens CL. Role of the vitreous in idiopathic preretinal macular fibrosis. Am J Ophthalmol. 1986 Feb 15;101(2):166-9. doi: 10.1016/0002-9394(86)90589-1. PMID 3946531
- [Background] Wise GN. Relationship of idiopathic preretinal macular fibrosis to posterior vitreous detachment. Am J Ophthalmol. 1975 Mar;79(3):358-62. doi: 10.1016/0002-9394(75)90606-6. PMID 1121991
- [Background] Mitchell P, Smith W, Chey T, Wang JJ, Chang A. Prevalence and associations of epiretinal membranes. The Blue Mountains Eye Study, Australia. Ophthalmology. 1997 Jun;104(6):1033-40. doi: 10.1016/s0161-6420(97)30190-0. PMID 9186446
- [Background] Kawasaki R, Wang JJ, Sato H, Mitchell P, Kato T, Kawata S, Kayama T, Yamashita H, Wong TY. Prevalence and associations of epiretinal membranes in an adult Japanese population: the Funagata study. Eye (Lond). 2009 May;23(5):1045-51. doi: 10.1038/eye.2008.238. Epub 2008 Aug 8. PMID 19440207
- [Background] Smiddy WE, Maguire AM, Green WR, Michels RG, de la Cruz Z, Enger C, Jaeger M, Rice TA. Idiopathic epiretinal membranes. Ultrastructural characteristics and clinicopathologic correlation. Ophthalmology. 1989 Jun;96(6):811-20; discussion 821. doi: 10.1016/s0161-6420(89)32811-9. PMID 2740079
- [Background] Wiznia RA. Posterior vitreous detachment and idiopathic preretinal macular gliosis. Am J Ophthalmol. 1986 Aug 15;102(2):196-8. doi: 10.1016/0002-9394(86)90144-3. PMID 3740180
- [Background] Sidd RJ, Fine SL, Owens SL, Patz A. Idiopathic preretinal gliosis. Am J Ophthalmol. 1982 Jul;94(1):44-8. doi: 10.1016/0002-9394(82)90189-1. PMID 7091281
- [Background] Bellhorn MB, Friedman AH, Wise GN, Henkind P. Ultrastructure and clinicopathologic correlation of idiopathic preretinal macular fibrosis. Am J Ophthalmol. 1975 Mar;79(3):366-73. doi: 10.1016/0002-9394(75)90608-x. PMID 1121993
- [Background] Clarkson JG, Green WR, Massof D. A histopathologic review of 168 cases of preretinal membrane. 1977. Retina. 2005 Jul-Aug;25(5 Suppl):1-17. doi: 10.1097/00006982-200507001-00006. No abstract available. PMID 16049358
- [Background] Appiah AP, Hirose T, Kado M. A review of 324 cases of idiopathic premacular gliosis. Am J Ophthalmol. 1988 Nov 15;106(5):533-5. doi: 10.1016/0002-9394(88)90581-8. PMID 3189467
- [Background] Ting FS, Kwok AK. Treatment of epiretinal membrane: an update. Hong Kong Med J. 2005 Dec;11(6):496-502. PMID 16340027
- [Background] Michels RG. A clinical and histopathologic study of epiretinal membranes affecting the macula and removed by vitreous surgery. Trans Am Ophthalmol Soc. 1982;80:580-656. No abstract available. PMID 6763804
- [Background] Puliafito CA, Hee MR, Lin CP, Reichel E, Schuman JS, Duker JS, Izatt JA, Swanson EA, Fujimoto JG. Imaging of macular diseases with optical coherence tomography. Ophthalmology. 1995 Feb;102(2):217-29. doi: 10.1016/s0161-6420(95)31032-9. PMID 7862410
- [Background] Falkner-Radler CI, Glittenberg C, Hagen S, Benesch T, Binder S. Spectral-domain optical coherence tomography for monitoring epiretinal membrane surgery. Ophthalmology. 2010 Apr;117(4):798-805. doi: 10.1016/j.ophtha.2009.08.034. Epub 2010 Jan 4. PMID 20045567
- [Background] Fraser-Bell S, Guzowski M, Rochtchina E, Wang JJ, Mitchell P. Five-year cumulative incidence and progression of epiretinal membranes: the Blue Mountains Eye Study. Ophthalmology. 2003 Jan;110(1):34-40. doi: 10.1016/s0161-6420(02)01443-4. PMID 12511343
- [Background] Kwok AKh, Lai TY, Yuen KS. Epiretinal membrane surgery with or without internal limiting membrane peeling. Clin Exp Ophthalmol. 2005 Aug;33(4):379-85. doi: 10.1111/j.1442-9071.2005.01015.x. PMID 16033350
- [Background] Grewing R, Mester U. Results of surgery for epiretinal membranes and their recurrences. Br J Ophthalmol. 1996 Apr;80(4):323-6. doi: 10.1136/bjo.80.4.323. PMID 8703883
- [Background] Park DW, Dugel PU, Garda J, Sipperley JO, Thach A, Sneed SR, Blaisdell J. Macular pucker removal with and without internal limiting membrane peeling: pilot study. Ophthalmology. 2003 Jan;110(1):62-4. doi: 10.1016/s0161-6420(02)01440-9. PMID 12511347
- [Background] Bovey EH, Uffer S, Achache F. Surgery for epimacular membrane: impact of retinal internal limiting membrane removal on functional outcome. Retina. 2004 Oct;24(5):728-35. doi: 10.1097/00006982-200410000-00007. PMID 15492626
- [Background] Burk SE, Da Mata AP, Snyder ME, Rosa RH Jr, Foster RE. Indocyanine green-assisted peeling of the retinal internal limiting membrane. Ophthalmology. 2000 Nov;107(11):2010-4. doi: 10.1016/s0161-6420(00)00375-4. PMID 11054324
- [Background] Gale JS, Proulx AA, Gonder JR, Mao AJ, Hutnik CM. Comparison of the in vitro toxicity of indocyanine green to that of trypan blue in human retinal pigment epithelium cell cultures. Am J Ophthalmol. 2004 Jul;138(1):64-9. doi: 10.1016/j.ajo.2004.02.061. PMID 15234283
- [Background] Yuen D, Gonder J, Proulx A, Liu H, Hutnik C. Comparison of the in vitro safety of intraocular dyes using two retinal cell lines: a focus on brilliant blue G and indocyanine green. Am J Ophthalmol. 2009 Feb;147(2):251-259.e2. doi: 10.1016/j.ajo.2008.08.031. Epub 2008 Nov 7. PMID 18992870
- [Background] Lim JW, Kim HK, Cho DY. Macular function and ultrastructure of the internal limiting membrane removed during surgery for idiopathic epiretinal membrane. Clin Exp Ophthalmol. 2011 Jan;39(1):9-14. doi: 10.1111/j.1442-9071.2010.02377.x. PMID 20662848
- [Background] Lee JW, Kim IT. Outcomes of idiopathic macular epiretinal membrane removal with and without internal limiting membrane peeling: a comparative study. Jpn J Ophthalmol. 2010 Mar;54(2):129-34. doi: 10.1007/s10384-009-0778-0. Epub 2010 Apr 18. PMID 20401561